CLINICAL TRIAL: NCT00647114
Title: A Phase I Study to Evaluate the Safety/Tolerability and Immunogenicity of V930/V932 in Patients With Cancer Expressing HER-2 and/or CEA
Brief Title: A Study to Test V930/V932 in Patients With Cancers Expressing Human Epidermal Growth Factor Receptor 2 (HER-2) and/or Carcinoembryonic Antigen (CEA)(V930-003)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Executive Vice President, Clinical and Quantitative Sciences, Merck & Co., Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V930-003; 2007_671
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Cancer
Keywords: Cancers expressing HER-2 and/or CEA
MeSH Terms: conditions — Neoplasms

ARMS (2):
- 1 (Experimental): V930
  Interventions: Biological: V930
- 2 (Experimental): V932
  Interventions: Biological: V932

INTERVENTIONS:
Biological: V930 — V930 - Over a 94 week duration, patients will receive a series of 5 injections (2.5 mg/injection), one every other week. Within 2 minutes of each injection of V930, each patient will be given an EP-IM injection consisting of two 60 msec pulses.
  Arms: 1
Biological: V932 — V932 - Over a 94 week duration, patients will receive a series of 5 injections, 6 patients will initially received intramuscular V932 vaccinations at a low dose (0.5x109 vg/injection),and following a safety assessment, up to an additional 35 patients will be treated with the high dose V932 (0.5x1011 vg/injection).
  Arms: 2

SUMMARY:
Treatment of patients with cancer types known to express the HER-2 and/or CEA tumor antigens.

DETAILED DESCRIPTION:
The optional followup period for this study is 1 year after the last vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have completed surgical treatment for his/her primary disease at least 1 month prior to enrollment
* Patient must not be pregnant 3 days prior to enrollment

Exclusion Criteria:

* Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of signing informed consent
* Patient has had their spleen removed or has a history of autoimmune disorders
* Patient is a regular user of any illicit drugs or has used within the past year of drug or alcohol abuse
* Patient is pregnant or breastfeeding or is expecting to conceive anytime following the study
* Patient is known to be Human Immunodeficiency Virus (HIV)-seropositive
* Patient has a known history of Hepatitis B or C
* Patient has received a vaccine for any disease or condition within one month of enrollment
* Patient has a primary central nervous system tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of V930/V932 followed by EP in cancer patients | Week 22

SECONDARY OUTCOMES:
To determine whether V930/V932 can elicit HER-2 specific and CEA specific immune responses measured using an ELISPOT assay | Week 22

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Diaz CM, Chiappori A, Aurisicchio L, Bagchi A, Clark J, Dubey S, Fridman A, Fabregas JC, Marshall J, Scarselli E, La Monica N, Ciliberto G, Montero AJ. Phase 1 studies of the safety and immunogenicity of electroporated HER2/CEA DNA vaccine followed by adenoviral boost immunization in patients with solid tumors. J Transl Med. 2013 Mar 8;11:62. doi: 10.1186/1479-5876-11-62. PMID 23497415